CLINICAL TRIAL: NCT03308682
Title: Safety and Dosimetry of a Long-lasting Radiolabeled Somatostatin Analogue 177Lu-DOTA-EB-TATE in Patients With Advanced Metastatic Neuroendocrine Tumors
Brief Title: 177Lu-DOTA-EB-TATE in Patients With Advanced Neuroendocrine Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-EB-3; ZIAEB000073 (NIH)
Record Dates: First submitted 2017-10-08; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-05

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — (177)Lu-DOTA-EB-TATE

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-DOTA-EB-TATE dosimetry calculation (Experimental): The patients were intravenously injected with single dose 0.50GBq-0.70GBq (13.5-18.9 mCi) of 177Lu-DOTA-EB-TATE and monitored at 2, 24, 72, 120 and 168 hours post-injection.
  Interventions: Drug: 177Lu-DOTA-EB-TATE

INTERVENTIONS:
Drug: 177Lu-DOTA-EB-TATE — The patients were intravenously injected with single dose 0.50GBq-0.70GBq (13.5-18.9 mCi) of 177Lu-DOTA-EB-TATE and monitored at 2, 24, 72, 120 and 168 hours post-injection.

SUMMARY:
This is an open-label, non-controlled, non-randomized study to investigate the long-lasting radiolabeled somatostatin analogue based peptide receptor radionuclide therapy and evaluation safety and dosimetry of 177Lu-DOTA-EB-TATE in patients with advanced metastatic neuroendocrine tumors. A single dose of 0.50GBq-0.70GBq (13.5-18.9 mCi) of 177Lu-DOTA-EB-TATE will be injected intravenously. and monitored at 2, 24, 72,120 and 168 hours post-injection with semiquantitative method based on quantitative single-photon emission computed tomography/computed tomography (SPECT/CT) performance.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NETs) are a heterogeneous group of neoplasms that can develop anywhere in the body and arise from neuroendocrine cells throughout the endocrine system. The most recent NCCN guidelines for unresectable and metastatic NET recommend somatostatin analogues as first-line treatment, but do not recommend a particular treatment sequence for the remaining therapies. Radiolabeled somatostatin analogue therapy, also known as peptide receptor radionuclide therapy has become a well-accepted treatment for patients with well to moderately differentiated unresectable or metastatic NETs and disease progression after first-line treatment. However, a major problem in the therapeutic use of 177Lu-Dotatate has been its short half-life and fast rate of clearance. This study was designed to investigate the safety, dosimetry and preliminary effects of a long-lasting radiolabeled somatostatin analogue 177Lu-DOTA-EB-TATE in patients with advanced metastatic neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* Adults who had neuroendocrine tumors and had metastasized, that were with histologically confirmed, inoperable and had showed disease progression according to Response Evaluation Criteria in Solid Tumors [RECIST]. Tumors were with well-differentiated histologic features and a Ki67 index of 0 to 20%. Target tumors were selected from CT, MRI, and 68Ga-DOTA-TATE PET/CT, with confirmed somatostatin receptor-expressing and at least one lesion has higher uptake than that of normal liver parenchyma on 68Ga-DOTA-TATE PET imaging within 1 weeks.

Exclusion Criteria:

* The exclusion criteria were a serum creatinine level of more than 150 μmol per liter, baseline measured GFR of less than 50 mL/min/1.73 m2, determined by 99mTc-DTPA renal function examination, a hemoglobin level of less than 8.0 g/dl, a white-cell count of less than 2.0× 109/L, a platelet count of less than 75 × 109/L, a total bilirubin level of more than 3 times the upper limit of the normal range and a serum albumin level of more than 3.0 g per deciliter, cardiac insufficiency including carcinoid heart valve disease, a severe allergy or hypersensitivity to radiographic contrast material, claustrophobia, and pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 177Lu-DOTA-EB-TATE in normal organs and metastatic neuroendocrine Tumors | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value at each time point in normal organs and metastatic neuroendocrine tumors will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 2 months
  Adverse events within 2 months after the injection and scanning of patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, M.D.,PhD., Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China